CLINICAL TRIAL: NCT02953340
Title: Randomized, OpEn-Label, Active-ContrOl Trial of SPI-2012 (Eflapegrastim) Versus Pegfilgrastim in the Management of Chemotherapy-Induced Neutropenia in Early-Stage BReast Cancer Patients Receiving Docetaxel and Cyclophosphamide (TC) (RECOVER)
Brief Title: SPI-2012 vs Pegfilgrastim in Management of Neutropenia in Breast Cancer Participants With Docetaxel and Cyclophosphamide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPI-GCF-302; 2016-003469-24 (EudraCT Number)
Record Dates: First submitted 2016-10-27; First posted 2016-11-02 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-01

CONDITIONS: Neutropenia; Breast Cancer
Keywords: Neutropenia; Breast Cancer; Long-acting Granulocyte Colony Stimulating Factor; Early Stage Breast Cancer; Docetaxel + Cyclophosphamide (TC) chemotherapy
MeSH Terms: conditions — Neutropenia; Breast Neoplasms | interventions — eflapegrastim; pegfilgrastim; Docetaxel; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- (Arm 1): SPI-2012 and TC (Experimental): At each cycle for 4 cycles, participants received SPI-2012 at a fixed dose of 13.2 milligrams (mg)/0.6 milliliter (mL), [3.6 mg granulocyte colony-stimulating factor {G-CSF}] subcutaneously (SC) approximately 24-26 hours after receiving intravenous (IV) infusion of docetaxel 75 mg/m^2 and cyclophosphamide 600 mg/m^2 IV infusion per institute's standard of care. All participants were followed for 35 (±5) days after last study treatment or patient discontinuation and long-term safety follow-up continued for 12 months after last dose of study treatment.
  Interventions: Drug: SPI-2012; Drug: Docetaxel; Drug: Cyclophosphamide
- (Arm 2): Pegfilgrastim and TC (Experimental): At each cycle for 4 cycles, participants received pegfilgrastim 6 mg (6 mg/0.6 mL GCSF) SC approximately 24-26 hours after receiving IV infusion of docetaxel 75 mg/m^2 and cyclophosphamide 600 mg/m^2 IV infusion per institute's standard of care. All participants were followed for 35 (±5) days after last study treatment or patient discontinuation and long-term safety follow-up continued for 12 months after last dose of study treatment.
  Interventions: Drug: Pegfilgrastim; Drug: Docetaxel; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: SPI-2012 — Supplied in prefilled single-use syringes for subcutaneous injection, administered on Day 2 of each cycle
  Other Names: HM10460A; Rolontis®; Eflapegrastim
  Arms: (Arm 1): SPI-2012 and TC
Drug: Pegfilgrastim — Subcutaneous injection administered on Day 2 of each cycle.
  Other Names: Neulasta®
  Arms: (Arm 2): Pegfilgrastim and TC
Drug: Docetaxel — 75mg/m^2 IV infusion administered on Day 1 of each cycle
  Other Names: Taxotere
Drug: Cyclophosphamide — 600mg/m^2 IV infusion administered on Day 1 of each cycle
  Other Names: Cytoxan

SUMMARY:
The purpose of this study is to compare the efficacy of SPI-2012 versus pegfilgrastim in participants with early-stage breast cancer receiving docetaxel and cyclophosphamide (TC) as measured by the duration of severe neutropenia (DSN).

DETAILED DESCRIPTION:
This is a Phase 3, randomized, open-label, active-controlled, multicenter study to compare the efficacy and safety of SPI-2012 versus pegfilgrastim in participants with early-stage breast cancer treated with TC chemotherapy as measured by the duration of severe neutropenia (DSN).

Each cycle was 21 days. Four cycles were evaluated for this study. On Day 1 of each cycle, participants received TC chemotherapy. On Day 2 of each cycle, participants received study drug (SPI-2012 or pegfilgrastim).

After cycle 1, as applicable, participants who received at least one dose of study drug will be followed for safety for 12 months after the last dose of study treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* New diagnosis of histologically confirmed early-stage breast cancer (ESBC), defined as operable Stage I to Stage IIIA breast cancer
* Candidate for adjuvant or neo-adjuvant TC chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status <= 2
* Absolute neutrophil count (ANC) >=1.5×10^9/L
* Platelet count >=100×10^9/L
* Hemoglobin >9 g/dL
* Calculated creatinine clearance > 50 mL/min
* Total bilirubin <=1.5 mg/dL
* Aspartate aminotransferase (AST) / Serum glutamic oxaloacetic transaminase (SGOT) and Alanine aminotransferase (ALT)/Serum glutamic pyruvic transaminase (SGPT) <=2.5×ULN (upper limit of normal)
* Alkaline phosphatase <=2.0×ULN

Key Exclusion Criteria:

* Active concurrent malignancy (except non melanoma skin cancer or carcinoma in situ of the cervix) or life-threatening disease
* Locally recurrent/metastatic breast cancer
* Known sensitivity to E. coli-derived products
* Concurrent adjuvant cancer therapy
* Previous exposure to filgrastim, pegfilgrastim, or other G-CSF products in clinical development within 12 months prior to the administration of study drug
* Active infection, receiving anti-infectives, or any underlying medical condition that would impair ability to receive protocol treatment
* Prior bone marrow or stem cell transplant
* Used any investigational drugs, biologics, or devices within 30 days prior to study treatment or plans to use any of these during the course of the study• Radiation therapy within 30 days prior to enrollment
* Major surgery within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2019-05-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (74):
- United States (49):
  - ACRC/ Arizona Clinical Research Center Inc., Tucson, Arizona
  - Yuma Regional Cancer Center, Yuma, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - NEA Baptist Clinic | Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Compassionate Care Research Group, Inc., Fountain Valley, California
  - California Cancer Associates for Research and Excellence Inc., Fresno, California
  - Pacific Shores Medical Group, Long Beach, California
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - Desert Regional Medical Center, Palm Springs, California
  - Emad Ibrahim, MD, INC., Redlands, California
  - Innovative Clinical Research Institute/ The Oncology Institute of Hope and Innovation, Whittier, California
  - Denver Health & Hospital Authority, Denver, Colorado
  - Pasco Pinellas Cancer Center, Holiday, Florida
  - Lakes Research, LLC, Miami Lakes, Florida
  - Mid-Florida Hematology and Oncology Centers, Orange City, Florida
  - Millennium Oncology, Pembroke Pines, Florida
  - BRCR Medical Center Inc, Plantation, Florida
  - Pinellas Hematology and Oncology, St. Petersburg, Florida
  - Bond & Steele Clinic, PA., Winter Haven, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Cancer Center of Middle Georgia, Dublin, Georgia
  - Dwight D. Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Oncology Specialists, SC, Park Ridge, Illinois
  - FPN Oncology and Hematology Specialists, Indianapolis, Indiana
  - Commonwealth Hematology-Oncology, PSC, Danville, Kentucky
  - Pontchartrain Cancer Center, Covington, Louisiana
  - Quest Research Institute, Royal Oak, Michigan
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - Freeman Health Systems, Joplin, Missouri
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - CHI Health St Francis, St Francis Cancer Treatment Center, Grand Island, Nebraska
  - Waverly Hematology Oncology, Cary, North Carolina
  - Gaston Hematology & Oncology Associates, PC, Gastonia, North Carolina
  - Aultman Hospital, Canton, Ohio
  - The Christ Hospital Cancer Center, Cincinnati, Ohio
  - St. Elizabeth Youngstown Hospital JACBCC/Oncology/ Mercy Health Youngstown LLC, Youngstown, Ohio
  - Carolina Blood and Cancer Care Associates, Rock Hill, South Carolina
  - The West Clinic, PC, d/b/a West Cancer Center, Germantown, Tennessee
  - CHI St Joseph Health Cancer Center, Bryan, Texas
  - Envision Cancer Center, LLC, Laredo, Texas
  - Texas Oncology, PA- McAllen South 2nd Street, McAllen, Texas
  - HOPE Cancer Center of East Texas, Tyler, Texas
  - Delta Hematology/Oncology Associates, Portsmouth, Virginia
  - Providence Regional Center Partnership, Everett, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - West Virginia University, Morgantown, West Virginia
- Canada (2):
  - CISSS de la Montérégie-Centre, Longueuil, Quebec
  - Jewish General Hospital, Montreal, Quebec
- Hungary (6):
  - Magyar Honvedseg Egeszsegugyi Kozpont, Onkologiai Osztaly, Budapest
  - Szent Imre Egyetemi Oktatokorhaz, Klinikai Onkologiai Osztaly, Budapest
  - Orszagos Onkologiai Intezet, ""B"" Belgyogyaszati Onkologiai Osztaly, Budapest
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Okato Korhaz, Klinikai Onkologiai es Sugarterapias Centrum, Miskolc
  - Szabolcs-Szatmar-Bereg Megyei Korhazak, Egyetemi Oktato Korhaz, Onkoradiologiai Osztaly, Nyíregyháza
  - Tolna Megyei Balassa Janos Korhaz, Klinikai Onkologiai Osztaly, Szekszárd
- India (2):
  - KEM Hospital Research Centre, Pune, Maharashtra
  - Christian Medical College, Vellore, Tamil Nadu
- Poland (7):
  - BIALOSTOCKIE CENTRUM ONKOLOGII im. Marii Sklodowskiej-Curie Oddzial Onkologii Klinicznej im. Ewy Pileckiej z Pododdzialem Chemioterapii dziennej, Bialystok
  - Regionalny Szpital Specjalistyczny im. dr Wladyslawa Bieganskiego Oddział Onkologii Klinicznej, Grudziądz
  - Instytut Centrum Zdrowia Matki Polki Klinika Chirurgii Onkologicznej i Chorob Piersi z Pododdzialem Onkologii Klinicznej, Lodz
  - Pracownia Leku Cytotoksycznego Szpitala Klinicznego Przemienienia Panskiego UM im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Szpital Rejonowy im. Dr. Jozefa Rostka w Raciborzu Dzienny Oddzial Chemioterapii, Racibórz
  - MrukMed. Lekarz Beata Madej Mruk i Partner. Spolka Partnerska Oddzial nr 1 w Rzeszowie, Rzeszów
  - Zachodniopomorskie Centrum Onkologii Osrodek Innowacyjnosci, Rozwoju i Badan Klinicznych, Szczecin
- South Korea (8):
  - Samsung Medical Center, Irwon-ro, Gangnam-gu Seoul
  - Wonju Severance Christian Hospital, Ilsan-ro, Gangwon-do
  - National Cancer Center, IIsan-ro, Gyeonggi-do
  - Cha Bundang Medical Center, Yatap-ro, Gyeonggi-do
  - Seoul National University Hospital, Daehwa-ro, Jongno-gu Seoul
  - Inha University Hospital, Inhang-ro, Jung-guIncheon
  - Korea University Anam Hospital, Inchon-ro, Seongbuk-guSeoul
  - Severance Hospital, Yonsei-ro, Seoul

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 74 sites in the United States, Canada, Hungary, Poland, India, Korea from 10 May 2017 to 06 May 2019. The study was conducted in two periods: treatment period (first dose of TC until 35 (± 5) days after last dose of treatment) and safety follow-up period (End of Treatment Visit through 12 months after last dose of study treatment).
Pre-assignment Details: A total of 237 participants were randomized into study, 118 participants in Arm 1 (SPI-2012 and TC) and 119 participants in Arm 2 (Pegfilgrastim and TC). 235 participants were treated, out of which 181 participants completed the study. All participants who received at least one dose of study drug (treatment period) entered the safety follow-up period.
Period: Overall Study
Arm/Group | (Arm 1): SPI-2012 and TC | (Arm 2): Pegfilgrastim and TC
Started | 118 | 119
Safety Population (Safety Population includes all participants who receive at least one dose of any protocol-specified drug (TC, SPI-2012 or pegfilgrastim).) | 117 | 118
Entered Safety Follow-up Period (Safety Follow-up Period included all participants who received at least one dose of any protocol specified drug (TC or SPI-2012 or pegfilgrastim) and continued for 12 months after last study treatment.) | 117 | 118
Completed | 96 | 85
Not Completed | 22 | 34
Not completed — Death | 0 | 1
Not completed — Investigator Decision | 3 | 3
Not completed — Initiated Non-Protocol Therapy | 5 | 14
Not completed — Myeloid Growth Factors Treatment | 0 | 1
Not completed — Withdrawal by Subject | 9 | 9
Not completed — Sponsor decision | 0 | 2
Not completed — Lost to Follow-up | 3 | 2
Not completed — Reason not specified | 2 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population includes all participants who were randomized.
Groups:
- (Arm 1): SPI-2012 and TC: At each cycle for 4 cycles, participants received SPI-2012 at a fixed dose of 13.2 mg/0.6 mL, [3.6 mg granulocyte colony-stimulating factor {G-CSF}] SC approximately 24-26 hours after receiving IV infusion of docetaxel 75 mg/m^2 and cyclophosphamide 600 mg/m^2 IV infusion per institute's standard of care. All participants were followed for 35 (±5) days after last study treatment or patient discontinuation and long-term safety follow-up continued for 12 months after last dose of study treatment.
- (Arm 2): Pegfilgrastim and TC: At each cycle for 4 cycles, participants received pegfilgrastim 6 mg (6 mg/0.6 mL G-CSF) SC approximately 24-26 hours after receiving IV infusion of docetaxel 75 mg/m^2 and cyclophosphamide 600 mg/m^2 IV infusion per institute's standard of care. All participants were followed for 35 (±5) days after last study treatment or patient discontinuation and long-term safety follow-up continued for 12 months after last dose of study treatment.
- Total: Total of all reporting groups
Arm/Group | (Arm 1): SPI-2012 and TC | (Arm 2): Pegfilgrastim and TC | Total
Number analyzed (Participants) | 118 | 119 | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (11.27) | 58.1 (12.67) | 58.0 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 119 | 237
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 15 | 33
  Not Hispanic or Latino | 100 | 104 | 204
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 85 | 96 | 181
  Black or African American | 11 | 7 | 18
  Asian | 20 | 16 | 36
  American Indian or Alaska Native | 1 | 0 | 1
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Duration of Severe Neutropenia (DSN) in Cycle 1
Description: DSN was defined as the number of days of severe neutropenia (absolute neutrophil count [ANC] <0.5×10^9 per liter [L]) from the first occurrence of ANC below the threshold.
Time Frame: Day 1 and daily on Days 4-15 in Cycle 1 (each cycle = 21 days)
Population: ITT population included all participants who were randomized.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | (Arm 1): SPI-2012 and TC | (Arm 2): Pegfilgrastim and TC
Number analyzed (Participants) | 118 | 119
Days | 0.31 (0.688) | 0.39 (0.949)
Statistical Analysis 1: Comparison: (Arm 1): SPI-2012 and TC vs (Arm 2): Pegfilgrastim and TC; Test type: Non-Inferiority — The study used non inferiority margin of 0.62 days for the above comparison. The non-inferiority of SPI-2012 to Pegfilgrastim was declared if the upper bound of 95% confidence interval (CI) of the difference in mean DSN between the treatment arms was <0.62 days; p < 0.0001, t-statistics; The p-values are based on the calculated t-statistics from the bootstrapped sample mean and standard deviation; Mean difference = -0.074, 95% CI 2-sided [-0.292 to 0.129]

2. Secondary Outcome: Time to Absolute Neutrophil Count (ANC) Recovery in Cycle 1
Description: Time to ANC recovery was defined as the time from chemotherapy administration until the participants ANC increased to >=1.5×10^9/L after the expected nadir. For participants with ANC value >=1.5×10^9/L at all times, time to ANC Recovery was assigned a value of 0.
Time Frame: Day 1 and daily on Days 4-15 in Cycle 1 (each cycle = 21 days)
Population: ITT population included all participants who were randomized.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | (Arm 1): SPI-2012 and TC | (Arm 2): Pegfilgrastim and TC
Number analyzed (Participants) | 118 | 119
Days | 3.49 (3.723) | 3.35 (3.745)

3. Secondary Outcome: Depth of ANC Nadir in Cycle 1
Description: The depth of ANC Nadir was defined as the lowest ANC value after administration of study drug (SPI-2012 or pegfilgrastim) in Cycle 1.
Time Frame: Day 1 and daily on Days 4-15 in Cycle 1 (each cycle = 21 days)
Population: ITT population included all participants who were randomized. Here 'N' (number of participants analyzed) signifies the number of participants evaluable for this outcome measure at the specified timepoint.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | (Arm 1): SPI-2012 and TC | (Arm 2): Pegfilgrastim and TC
Number analyzed (Participants) | 115 | 116
10^9 cells/L | 2.67 (3.504) | 2.06 (2.034)

4. Secondary Outcome: Number of Participants With Febrile Neutropenia (FN) in Cycle 1
Description: FN was defined as an oral temperature >38.3 degree Celsius (°C) (101.0 degrees Fahrenheit [°F]) or two consecutive readings of >38.0°C (100.4°F) for 2 hours and ANC <1.0×10^9/L.
Time Frame: Day 1 and daily on Days 4-15 in Cycle 1 (each cycle = 21 days)
Population: ITT population included all participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | (Arm 1): SPI-2012 and TC | (Arm 2): Pegfilgrastim and TC
Number analyzed (Participants) | 118 | 119
Participants | 1 | 4

5. Secondary Outcome: Duration of Severe Neutropenia (DSN) in Cycles 2, 3 and 4
Description: DSN was defined as the number of days of severe neutropenia (ANC <0.5×10^9/L) from the first occurrence of ANC below the threshold.
Time Frame: Days 1, 4, 7, 10, and 15 of Cycles 2, 3, and 4 (each cycle = 21 days)
Population: ITT population included all participants who were randomized.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | (Arm 1): SPI-2012 and TC | (Arm 2): Pegfilgrastim and TC
Number analyzed (Participants) | 118 | 119
Days
  Cycle 2 | 0.08 (0.267) | 0.09 (0.432)
  Cycle 3 | 0.07 (0.252) | 0.07 (0.283)
  Cycle 4 | 0.07 (0.252) | 0.08 (0.266)

6. Secondary Outcome: Number of Participants With Neutropenic Complications in Cycle 1
Description: Neutropenic complications refer to hospitalizations due to neutropenic events and/or the use of anti-infectives due to neutropenia.
Time Frame: Day 1 and daily on Days 4-15 in Cycle 1 (each cycle = 21 days)
Population: ITT population included all participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | (Arm 1): SPI-2012 and TC | (Arm 2): Pegfilgrastim and TC
Number analyzed (Participants) | 118 | 119
Participants | 1 | 5

7. Secondary Outcome: Number of Participants With Febrile Neutropenia in Cycles 2, 3 and 4
Description: FN was defined as an oral temperature >38.3°C (101.0°F) or two consecutive readings of >38.0°C (100.4°F) for 2 hours and ANC <1.0×10^9/L.
Time Frame: Days 1, 4, 7, 10, and 15 of Cycles 2, 3, and 4 (each cycle = 21 days)
Population: ITT population included all participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | (Arm 1): SPI-2012 and TC | (Arm 2): Pegfilgrastim and TC
Number analyzed (Participants) | 118 | 119
Participants
  Cycle 2 | 0 | 2
  Cycle 3 | 0 | 0
  Cycle 4 | 0 | 0

8. Secondary Outcome: Relative Dose Intensity (RDI) of TC Chemotherapy
Description: RDI was defined as the percentage of the planned dose of TC chemotherapy that each participant actually received during the study, and is expressed as the total dose received, divided by total dose planned multiplied by 100. The planned dose was defined as the dose that would be given if no doses were missed and/or no dose reductions were made for the number of cycles started. The total planned dose was the sum of planned doses over all cycles.
Time Frame: Cycles 1, 2, 3 and 4 (each cycle = 21 days)
Population: Safety analysis (SAF) population included all participants who received at least one dose of any protocol-specified drug (TC or SPI-2012 or pegfilgrastim).
Measure: Mean (Standard Deviation); unit: Percentage of planned dose
Arm/Group | (Arm 1): SPI-2012 and TC | (Arm 2): Pegfilgrastim and TC
Number analyzed (Participants) | 117 | 118
Percentage of planned dose
  Docetaxel | 96.9 (7.70) | 98.4 (7.89)
  Cyclophosphamide | 98.4 (5.27) | 98.8 (6.40)

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs), and Death
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product or study procedure, whether or not considered related to the medicinal product. A TEAE is any AE that occurred from the first dose of study treatment through 12 months after the last dose of study treatment or 35 (±5) days after date of participant early discontinuation. SAE is defined as any AE which meets any of the following criteria: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in a persistent or significant disability/incapacity, results in a congenital anomaly/birth defect, includes important medical events.
Time Frame: Up to 4 cycles (each cycle = 21 days) plus a 12-month follow-up from the last dose (up to 15 months)
Population: SAF population included all participants who received at least one dose of any protocol-specified drug (TC or SPI-2012 or pegfilgrastim). Data was summarized and reported for Treatment and Follow-up period separately for both groups.
Measure: Count of Participants; unit: Participants
Groups:
- (Arm 1): SPI-2012 and TC: At each cycle for 4 cycles, participants received SPI-2012 at a fixed dose of 13.2 mg/0.6 mL, [3.6 mg granulocyte colony-stimulating factor {G-CSF}] SC approximately 24-26 hours after receiving IV infusion of docetaxel 75 mg/m^2 and cyclophosphamide 600 mg/m^2 IV infusion per institute's standard of care. All participants were followed for 35 (±5) days after last study treatment or patient discontinuation.
- (Arm 2): Pegfilgrastim and TC: At each cycle for 4 cycles, participants received pegfilgrastim 6 mg (6 mg/0.6 mL G-CSF) SC approximately 24-26 hours after receiving IV infusion of docetaxel 75 mg/m^2 and cyclophosphamide 600 mg/m^2 IV infusion per institute's standard of care. All participants were followed for 35 (±5) days after last study treatment or patient discontinuation.
- (Arm 1): SPI-2012 and TC: Follow-up Period; Arm 2: Pegfilgrastim and TC: Follow-up Period: In addition to the treatment period, long-term safety follow-up continued for 12 months after last study treatment.
Arm/Group | (Arm 1): SPI-2012 and TC | (Arm 2): Pegfilgrastim and TC | (Arm 1): SPI-2012 and TC: Follow-up Period | Arm 2: Pegfilgrastim and TC: Follow-up Period
Number analyzed (Participants) | 117 | 118 | 117 | 118
Participants
  TEAEs | 115 | 116 | 33 | 48
  SAEs | 12 | 19 | 2 | 4
  Death | 0 | 1 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: The number of participants with clinically significant hematology (including basophils, basophils/leukocytes, eosinophils, eosinophils/leukocytes, hematocrit, hemoglobin, lymphocytes, lymphocytes/leukocytes, monocytes, monocytes/leukocytes, neutrophils, neutrophils/leukocytes, platelets, and white blood cells) and serum chemistry (including alanine aminotransferase [ALT], alkaline phosphatase [ALP], aspartate aminotransferase [AST], bilirubin, calcium, cholesterol, creatinine, potassium, sodium, and triglycerides) laboratory abnormalities were reported. Clinically significant findings in laboratory parameters were based on investigator's discretion according to Common Technical Criteria for Adverse Events (CTCAE) Version 4.03.
Time Frame: Up to 4 cycles (each cycle = 21 days) plus a 12-month follow-up from the last dose (up to 15 months)
Population: SAF population included all participants who received at least one dose of any protocol-specified drug (TC or SPI-2012 or pegfilgrastim).
Measure: Count of Participants; unit: Participants
Arm/Group | (Arm 1): SPI-2012 and TC | (Arm 2): Pegfilgrastim and TC
Number analyzed (Participants) | 117 | 118
Participants
  Hematology: Basophils | 0 | 0
  Hematology: Basophils/Leukocytes | 0 | 0
  Hematology: Eosinophils | 0 | 0
  Hematology: Eosinophils/Leukocytes | 0 | 0
  Hematology: Hematocrit | 4 | 2
  Hematology: Hemoglobin | 6 | 4
  Hematology: Lymphocytes | 0 | 0
  Hematology: Lymphocytes/Leukocytes | 6 | 13
  Hematology: Monocytes | 0 | 0
  Hematology: Monocytes/Leukocytes | 0 | 0
  Hematology: Neutrophils | 17 | 23
  Hematology: Neutrophils/Leukocytes | 12 | 9
  Hematology: Platelets | 10 | 2
  Hematology: White Blood Cells | 16 | 18
  Chemistry: Alanine aminotransferase | 2 | 1
  Chemistry: Alkaline phosphatase | 0 | 1
  Chemistry: Aspartate aminotransferase | 1 | 1
  Chemistry: Bilirubin | 0 | 0
  Chemistry: Calcium | 1 | 1
  Chemistry: Cholesterol | 0 | 0
  Chemistry: Creatinine | 0 | 0
  Chemistry: Potassium | 0 | 1
  Chemistry: Sodium | 0 | 2
  Chemistry: Triglycerides | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 4 cycles (each cycle = 21 days) plus a 12-month follow-up from the last dose (up to 15 months)
Description: The Safety Analysis Population included all participants who received at least one dose of any protocol-specified drug (TC or SPI-2012 or pegfilgrastim). Adverse events data was summarized and reported for Treatment and Follow-up period separately for both groups.
Groups:
- (Arm 1): SPI-2012 and TC: At each cycle for 4 cycles, participants received SPI-2012 at a fixed dose of 13.2 mg / 0.6 mL, [3.6 mg G-CSF] SC approximately 24-26 hours after receiving IV infusion of docetaxel 75 mg/m^2 and cyclophosphamide 600 mg/m^2 IV infusion per institute's standard of care. All participants were followed for 35 (±5) days after the last study treatment or patient discontinuation.
- (Arm 2): Pegfilgrastim and TC: At each cycle for 4 cycles, participants received pegfilgrastim 6 mg (6 mg/0.6 mL G-CSF) SC approximately 24-26 hours after receiving IV infusion of docetaxel 75 mg/m^2 and cyclophosphamide 600 mg/m^2 IV infusion per institute's standard of care. All participants were followed for 35 (±5) days after the last study treatment or patient discontinuation.
- (Arm 2): Pegfilgrastim and TC: Follow-up Period: In addition to the treatment period, long-term safety follow-up continued for 12 months after last study treatment.
Arm/Group | (Arm 1): SPI-2012 and TC | (Arm 2): Pegfilgrastim and TC | (Arm 1): SPI-2012 and TC: Follow-up Period | (Arm 2): Pegfilgrastim and TC: Follow-up Period
All-Cause Mortality (participants affected / at risk) | 0/117 | 1/118 | 0/117 | 0/118
Serious Adverse Events (participants affected / at risk) | 12/117 | 19/118 | 2/117 | 4/118
Other Adverse Events (participants affected / at risk) | 115/117 | 116/118 | 33/117 | 48/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | (Arm 1): SPI-2012 and TC (N=117) | (Arm 2): Pegfilgrastim and TC (N=118) | (Arm 1): SPI-2012 and TC: Follow-up Period (N=117) | (Arm 2): Pegfilgrastim and TC: Follow-up Period (N=118)
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Administration site reaction (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Chest wall abscess (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | (Arm 1): SPI-2012 and TC (N=117) | (Arm 2): Pegfilgrastim and TC (N=118) | (Arm 1): SPI-2012 and TC: Follow-up Period (N=117) | (Arm 2): Pegfilgrastim and TC: Follow-up Period (N=118)
Flushing (Vascular disorders) | 9 | 10 | 0 | 2
Hot flush (Vascular disorders) | 10 | 8 | 1 | 3
Hypertension (Vascular disorders) | 4 | 8 | 1 | 3
Hypotension (Vascular disorders) | 6 | 3 | 0 | 0
Fatigue (General disorders) | 40 | 51 | 0 | 0
Pyrexia (General disorders) | 25 | 26 | 1 | 0
Oedema peripheral (General disorders) | 12 | 15 | 2 | 2
Asthenia (General disorders) | 15 | 11 | 0 | 0
Pain (General disorders) | 5 | 11 | 0 | 1
Chills (General disorders) | 4 | 6 | 0 | 1
Malaise (General disorders) | 3 | 6 | 0 | 0
Insomnia (Psychiatric disorders) | 18 | 11 | 1 | 1
Anxiety (Psychiatric disorders) | 5 | 8 | 0 | 0
Lymphocyte count decreased (Investigations) | 44 | 54 | 0 | 1
White blood cell count decreased (Investigations) | 22 | 31 | 1 | 2
Neutrophil count decreased (Investigations) | 16 | 22 | 1 | 0
Platelet count decreased (Investigations) | 12 | 3 | 0 | 0
White blood cell count increased (Investigations) | 9 | 3 | 0 | 0
Tachycardia (Cardiac disorders) | 5 | 6 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 37 | 37 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 22 | 11 | 1 | 2
Lymphopenia (Blood and lymphatic system disorders) | 10 | 9 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 17 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 14 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 10 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 0 | 0
Headache (Nervous system disorders) | 31 | 35 | 0 | 1
Dysgeusia (Nervous system disorders) | 9 | 16 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 9 | 14 | 1 | 1
Dizziness (Nervous system disorders) | 6 | 12 | 1 | 1
Lacrimation increased (Eye disorders) | 2 | 7 | 0 | 1
Nausea (Gastrointestinal disorders) | 50 | 61 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 38 | 40 | 1 | 3
Constipation (Gastrointestinal disorders) | 26 | 24 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 14 | 20 | 0 | 2
Vomiting (Gastrointestinal disorders) | 14 | 19 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 14 | 9 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 9 | 10 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 9 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 40 | 43 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 13 | 11 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 9 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 4 | 6 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 47 | 51 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 26 | 23 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 15 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 12 | 4 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 11 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 23 | 19 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 8 | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 8 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 9 | 1 | 2
Nasopharyngitis (Infections and infestations) | 3 | 6 | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 7 | 0 | 3
Candida infection (Infections and infestations) | 1 | 7 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-07-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT02953340/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT02953340/SAP_001.pdf